CLINICAL TRIAL: NCT06664632
Title: Effectiveness of Knee Sync Partner and Strengthening Exercises Versus Strengthening Exercises in Knee Osteoarthritis. A Randomized Controlled Trial.
Brief Title: Effectiveness of Knee Sync Partner and Strengthening Exercises Versus Strengthening Exercises in Knee Osteoarthritis.RCT
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Superior University (Other)
Responsible Party: Principal Investigator, Muhammad Naveed Babur, Principal Investigator, Superior University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: MSRSW/Batch-Fall22/745
Record Dates: First submitted 2024-10-28; First posted 2024-10-29 (Actual); Last update posted 2024-10-29 (Actual); Status verified 2024-10

CONDITIONS: Knee Osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exp Group (Experimental)
  Interventions: Behavioral: Exp
- Control Group (Active Comparator)
  Interventions: Diagnostic Test: control

INTERVENTIONS:
Behavioral: Exp — Participants in this group will receive treatment using the Knee Sync Partner, a novel portable device designed to provide electrical traction and stimulation specifically for the knee joint.
  controlled mechanical traction to the knee joint to reduce joint contact pressure, enhance synovial fluid flow, and increase joint space. This is expected to alleviate pain and improve mobility.
  Arms: Exp Group
Diagnostic Test: control — This will include a combination of isometric and isotonic exercises aimed at strengthening the knee musculature, enhancing joint stability, and reducing pain. The exercise regimen will focus on major muscle groups supporting the knee, such as the quadriceps, hamstrings, and calf muscles.
  Arms: Control Group

SUMMARY:
This study explores the effectiveness of a novel treatment approach for knee osteoarthritis (OA) by comparing the combined use of a new device, "Knee Sync Partner," which provides electrical knee traction with stimulation and strengthening exercises, to traditional strengthening exercises alone. Knee osteoarthritis is a leading cause of chronic pain and disability worldwide, significantly impacting the quality of life for many individuals, especially with the growing elderly population.

DETAILED DESCRIPTION:
While strengthening exercises are a well-established treatment for improving joint stability and mobility in knee OA patients, the potential benefits of integrating electrical stimulation and traction therapy remain underexplored. This research addresses the gap by conducting a randomized controlled trial to assess whether this combined approach leads to superior outcomes in terms of pain relief, functional improvement, and joint health. The findings could provide valuable insights into more effective, non-invasive management strategies for knee OA, expanding therapeutic options in physical therapy.

ELIGIBILITY:
Inclusion Criteria:

* having pain in knee for more than 3 months in most days of week
* age between 40 and 70 years
* patient who filled Kellgren-Lawrence radiographic criteria

Exclusion Criteria:

* joint injection in the previous three months.
* The exclusion criteria were patients who had inflammatory arthritis
* osteoarthritis of the hips.

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2023-11-01 (Actual); Primary Completion 2024-06-01 (Actual); Study Completion 2024-11-15 (Estimated)

PRIMARY OUTCOMES:
WOMAC Scale | 12 Months
  The scores for each subscale are summed up, with a possible score range of 0-20 for Pain, 0-8 for Stiffness, and 0-68 for Physical Function. Usually a sum of the scores for all three subscales gives a total WOMAC score

CONTACTS AND LOCATIONS:
Locations (1):
- Chaudary Muhammad Akram Teaching Hospital, Azra Naheed Medical College, Superior University, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No